CLINICAL TRIAL: NCT01500993
Title: 5-Fluorouracil Versus Capecitabine as Perioperative Treatment for Locally Advanced Rectal Cancer. a Randomized Phase III Trial
Brief Title: Capecitabine in the Perioperative Treatment of Rectal Cancer
Acronym: Rektum-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Frederik Wenz, Co-Investigator, Head Department of Radiation Oncology Mannheim, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rektum III
Record Dates: First submitted 2011-12-21; First posted 2011-12-29 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Chemoradiotherapy; Capecitabine; phase-III trial
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-Fluorouracil (5-FU) (Active Comparator): Drug - 5FU based chemoradiotherapy and chemotherapy
  Interventions: Drug: 5-FU
- Capecitabine (Experimental): Drug - Capecitabine-based radiochemotherapy and chemotherapy
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine standard therapy (i.e. 2,500 mg/sqm) x 5 cycles plus 1 cycle of capecitabine based chemoradiotherapy (1.650 mg/sqm)
  Other Names: Xeloda
  Arms: Capecitabine
Drug: 5-FU — 4 cycles of bolus 5-FU (500 mg/sqm) and 1 cycle of 5-FU based chemoradiotherapy (either 1,000 mg/sqm/day infusional 5-Fu days 1-5 and 29-33 or 225 mg/sqm/day infusional 5-Fu throughout the time of chemoradiotherapy)
  Other Names: 5-Fluorouracil
  Arms: 5-Fluorouracil (5-FU)

SUMMARY:
This study compares capecitabine with standard 5-FU in the perioperative treatment of locally advanced rectal cancer.

DETAILED DESCRIPTION:
5-Fluorouracil (5-FU) based chemoradiotherapy (CRT) is regarded a standard perioperative treatment in locally advanced rectal cancer (LARC). We investigate the replacement of 5-FU by the oral pro-drug capecitabine (cape) within a randomized phase III trial. Patients aged ≥18 years with LARC stage II or III are recruited into this two-arm, two-cohort randomized non-inferiority phase-III trial (arm A: cape, arm B: 5-FU; cohort [C] I: adjuvant, C II: neoadjuvant). Regimens: Arm A: CRT: 50.4 Gy + cape 1,650 mg/m² days 1-38 plus five cycles of cape 2,500 mg/m² d 1-14, repeated d 22 (C I: 2 x cape, CRT, 3 x cape; C II: CRT, TME surgery followed by cape x 5). Arm B: CRT: 50.4 Gy + infusional 5-FU 225 mg/m² daily [C I] or infusional 5-FU 1,000 mg/m² d 1-5 and 29-33 [C II] plus 4 cycles of bolus 5-FU 500mg/m² d 1-5, repeated d 29 (C I: 2 x 5-FU, CRT, 2 x 5-FU; C II: CRT, TME surgery followed by 5-FU x 4). Primary endpoint is 5-year overall survival (OS), secondary endpoints comprise 3-year disease-free survival (DFS) and safety.

The study is designed to investigate whether 5- year overall survival rate (SR5) is non-inferior in arm A versus arm B. We hypothesize that SR5 in the standard arm B is 57.5%. Sample size calculation is performed with a power of 80% and a type I error of 5% and with a drop-out rate of 5%. Therefore, a total of at least 372 evaluable patients (i.e. 186 per arm) is required to confirm non-inferiority of the experimental arm A with a non-inferiority margin of maximal 12.5% and a median follow-up time of 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are 18 years or older and have histologically confirmed adenocarcinoma of the rectum (defined as the distal border of the tumour less than 16 cm from the anal verge measured by rigid rectoscopy) with no evidence of distant metastases (identified by abdominal ultrasound or CT scan and chest radiography).
* Patients in the adjuvant cohort have undergone R0-resection by total mesorectal excision (TME) of a pT3-4 N any or T any N positive non-metastatic rectal cancer.
* Patients treated in the neoadjuvant cohort need to have a clinical T3-4 N any or T any N positive tumour staged by endoscopic ultrasound, provided the lower border of the tumour is located 0 - 16 cm from the anal verge measured by rigid rectoscopy and the primary tumour is deemed resectable by TME surgery on the basis of clinical assessment. Other eligibility criteria comprise: WHO status of zero or one; adequate liver, renal, and bone marrow function defined as follows: leucocyte count > 3,500/µl, thrombocyte count > 100,000/µl, hemoglobin > 10.0 g/dl; serum bilirubin < 2.0 mg/dl, serum creatinine < 2.0 mg/dl.

Exclusion criteria:

* Prior treatment for rectal cancer, prior chemo- or immunotherapy, prior pelvic radiotherapy, or a history of other malignant diseases within the past five years with the exception of successfully treated basal carcinoma of the skin or carcinoma in situ of the uterine cervix.
* Participation in another trial, pregnancy, breast-feeding, unwillingness to use effective contraception, or a medical condition or concomitant illness which could potentially interfere with compliance to the protocol are regarded as exclusion criteria, as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2002-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5-year

SECONDARY OUTCOMES:
disease-free survival (DFS) | 3-year DFS
Local recurrence rate | 5 years
  Percentage of patient with local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Hofheinz, MD, Study Chair — Universitätsmedizin Mannheim Germany, University of Heidelberg; Frederik Wenz, MD, Study Chair — Universitätsmedizin Mannheim, Germany, University of Heidelberg; Stefan Post, MD, Study Chair — Universitätsmedizin Mannheim, Germany, University of Heidelberg; Andreas Hochhaus, MD, Study Chair — Universitätsklinikum Jena, Germany
Locations (14):
- Germany (14):
  - Dr Martina Grunewald, Aschersleben
  - Dr Hans Walter Lindemann, Hagen
  - Prof Hartmut Link, Kaiserslautern
  - Dr Elisabeth Fritz, Koblenz
  - Dr Stephan Kremers, Lebach
  - Dr Lothar Müller, Leer
  - Dr Christain Constantin, Lemgo
  - Dr Erika Kettner, Magdeburg
  - Dr Markus Moehler, Mainz
  - Dr Udo Hieber, Mannheim
  - Prof Ralf Hofheinz, Mannheim
  - Dr Matthias Hipp, Regensburg
  - Prof Axel Matzdorff, Saarbrücken
  - Dr Stephan Laechelt, Tübingen

REFERENCES:
- [Result] Hofheinz RD, Wenz F, Post S, Matzdorff A, Laechelt S, Hartmann JT, Muller L, Link H, Moehler M, Kettner E, Fritz E, Hieber U, Lindemann HW, Grunewald M, Kremers S, Constantin C, Hipp M, Hartung G, Gencer D, Kienle P, Burkholder I, Hochhaus A. Chemoradiotherapy with capecitabine versus fluorouracil for locally advanced rectal cancer: a randomised, multicentre, non-inferiority, phase 3 trial. Lancet Oncol. 2012 Jun;13(6):579-88. doi: 10.1016/S1470-2045(12)70116-X. Epub 2012 Apr 13. PMID 22503032
- [Derived] Garcia-Albeniz X, Gallego R, Hofheinz RD, Fernandez-Esparrach G, Ayuso-Colella JR, Bombi JA, Conill C, Cuatrecasas M, Delgado S, Gines A, Miquel R, Pages M, Pineda E, Pereira V, Sosa A, Reig O, Victoria I, Feliz L, Maria de Lacy A, Castells A, Burkholder I, Hochhaus A, Maurel J. Adjuvant therapy sparing in rectal cancer achieving complete response after chemoradiation. World J Gastroenterol. 2014 Nov 14;20(42):15820-9. doi: 10.3748/wjg.v20.i42.15820. PMID 25400468